CLINICAL TRIAL: NCT07184983
Title: Telehealth-Delivered tDCS for Cannabis Addiction Recovery: The C.A.R.E.S. (Cannabis Addiction Recovery Enhancement Stimulation) Initiative
Brief Title: RS-tDCS for Cannabis Use Disorder: The C.A.R.E.S. Initiative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25-00489; 1UG3DA063344-01 (NIH)
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Cannabis Use Disorder
Keywords: Cannabis; CUD; tDCS; Transcranial Direct Current Stimulation; Neuromodulation; Brain Stimulation
MeSH Terms: conditions — Marijuana Abuse | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): Participants will complete 20 remotely supervised (RS) daily sessions, each 20 minutes, of active dorsolateral prefrontal cortex (DLPFC) tDCS combined with mindfulness meditation.
  Interventions: Device: Active Transcranial Direct Current Stimulation (tDCS); Behavioral: Mindfulness meditation
- Sham tDCS (Active Comparator): Participants will complete 20 RS sham sessions, each 20 minutes, of active DLPFC tDCS combined with mindfulness meditation.
  Interventions: Device: Sham Transcranial Direct Current Stimulation (tDCS); Behavioral: Mindfulness meditation

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation (tDCS) — tDCS is a noninvasive brain stimulation device that modulates brain activity by delivering low-intensity electrical current (2.0 mA) through scalp sponge electrodes. Device is programmed to ramp up to 2.0 mA (for 30 seconds), provide constant current throughout the session (19 minutes), and then ramp down (for 30 seconds) at the end.
  Arms: Active tDCS
Device: Sham Transcranial Direct Current Stimulation (tDCS) — tDCS is a noninvasive brain stimulation device that modulates brain activity by delivering low-intensity electrical current (2.0 mA) through scalp sponge electrodes. Device is programmed to ramp up to 2.0 mA (for 30 seconds) followed by a ramp down (30 seconds), with no current delivery for 18 minutes, and then ramp up (for 30 seconds) and down (for 30 seconds) at the end.
  Arms: Sham tDCS
Behavioral: Mindfulness meditation — Participants will follow an audio track for guided mindfulness during the stimulation.

SUMMARY:
The purpose of this sham-controlled pilot randomized controlled trial (RCT) is to evaluate the feasibility, safety, and preliminary efficacy of a one-month intervention consisting of 20 home-based active or sham RS-tDCS sessions paired with audio track guided mindfulness meditation practice in otherwise healthy adults seeking to reduce cannabis use in the context of cannabis use disorder (CUD).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 22-65 years (inclusive)
2. Currently meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for CUD, as determined by DSM-V criteria (M.I.N.I)
3. Positive for cannabis on the 11-COOH-THC single panel urine test
4. Seeking treatment to reduce or discontinue cannabis use (Marijuana Ladder ranged between 5-8 [inclusive])
5. Kessler Psychological Distress Scale (K10) score < 35 (minimal to moderate distress)
6. Wide Range Achievement Test-5(WRAT-5) score ≥ 85
7. Ability to use mobile devices
8. Fluent in English or Spanish

Exclusion Criteria:

1. Cannabis is used exclusively as prescribed or directed by their provider
2. Meets DSM-V criteria for substance use disorder within the past six months for any psychoactive substance other than cannabis
3. Meets DSM-V criteria for alcohol use disorder within the past six months
4. Primary psychiatric disorder (major depressive disorder, bipolar disorder, or psychotic disorder) as the principal diagnosis, independent of cannabis use disorder; or current diagnosis of bipolar disorder, psychotic disorder, or any other alcohol/substance use disorder as defined by DSM-5-TR and confirmed via the Mini-International Neuropsychiatric Interview (MINI).
5. Primary neurologic or major medical disorder that would interfere with study participation.
6. Enrolled in group or individual therapy for substance use disorder that would be concurrent with the study intervention
7. History of moderate or severe traumatic brain injury
8. Seizure disorder or recent (<5 years) seizure history
9. Presence of metal or active implants in the head/neck
10. Any skin disorder or skin sensitive area near stimulation locations
11. Pregnant or planning pregnancy during the study period or breastfeeding

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants who complete at least 70% (14 out of 20) of intervention sessions | End of treatment (up to 6 weeks)
The proportion of participants who discontinue due to adverse effects | End of treatment (up to 6 weeks)
The proportion of participants with no serious adverse events | End of treatment (up to 6 weeks)
Change in cannabis use frequency, measured by the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis-Use Inventory (DFAQ-CU) | Baseline, End of treatment (up to 6 weeks)
  The DFAQ-CU is a self-report scale used to assess cannabis use behaviors. It measures frequency, quantity, age of onset, and daily sessions of cannabis use, including different forms like dry product, concentrates, and edibles. The DFAQ-CU also includes visual aids and questions about methods of cannabis administration and tetrahydrocannabinol (THC) levels. Questions 2-3, 6-12 assess frequency.
Change in daily cannabis use, measured by the Timeline Followback (TLFB) method assessment | Baseline, End of treatment (up to 6 weeks)
  Daily cannabis use is assessed using the TLFB method, a validated self-report instrument used to collect retrospective estimates of daily cannabis use.
Change in cannabis withdrawal symptoms, measured by the Cannabis Withdrawal Scale (CWS) | Baseline, End of treatment (up to 6 weeks)
  The CWS assesses withdrawal symptoms experienced over the last 24 hours and consists of 19 statements. For each statement, its negative impact on normal daily activities is rated on a Likert scale from 0 (not at all) to 10 (extremely). The total score ranges from 0 to 190; higher scores indicate that withdrawal symptoms have a larger negative impact on normal daily activities.

SECONDARY OUTCOMES:
Change in cannabis craving, measured by the Marijuana Craving Questionnaire (MCQ-17) | Baseline, 1-month follow-up
Change in psychological distress as measured by the Kessler Psychological Distress Scale (K10) | Baseline, 1-month follow-up
  K10 is a 10-item questionnaire intended to yield a global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period. Each question is given a score between 1 (none of the time) to 5 (all of the time). The total score ranges from 10 to 50. People with scores < 20 are likely to be well, 20-24 are likely to have a mild mental disorder, 25-29 are likely to have moderate mental disorder, and > 30 are likely to have a severe mental disorder.
Change in anxiety as measured by State-Trait Anxiety Inventory (STAI) | Baseline, 1-month follow-up
  The STAI is a psychological tool used to measure both state anxiety (temporary feelings of nervousness) and trait anxiety (a general tendency to be anxious). It's a 40-item self-report questionnaire, 20 items allocated to each of the S-Anxiety and T-Anxiety subscales, that uses a 4-point Likert scale. Item scores are added to obtain subtest total scores. Scoring should be reversed for anxiety-absent items (19 items of the total 40). Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.
Change in function as measured by the Marijuana Problem Scale (MPS) | Baseline, 1-month follow-up
  The MPS (form AS5) is a self-report assessment that helps the patient identify areas their life affected by marijuana use. It contains 19 items that represent potential negative effects of marijuana on social relationships, self-esteem, motivation and productivity, work and finances, physical health, memory impairment, and legal problems. Items are rated either 0 (Not a problem), 1 (A minor problem), or 2 (A serious problem). Higher scores generally indicate more serious problems with marijuana.
Change in depression as measured by the Beck Depression Inventory (BDI) | Baseline, 1-month follow-up
  BDI is a 21-item self-report scale designed to measure the severity of depressive symptoms. Each item is scored 0-3. The total score range is 0-63; the higher the score, the more severe the depression. A score > 40 indicates extreme depression.
Change in cannabis use frequency, measured by the Daily Sessions, Frequency, Age of Onset, and Quantity of Cannabis-Use Inventory (DFAQ-CU) | Baseline, 1-month follow-up
  The DFAQ-CU is a self-report scale used to assess cannabis use behaviors. It measures frequency, quantity, age of onset, and daily sessions of cannabis use, including different forms like dry product, concentrates, and edibles. The DFAQ-CU also includes visual aids and questions about methods of cannabis administration and THC levels. Questions 2-3, 6-12 assess frequency.
Change in daily cannabis use, measured by the Timeline Followback Method Assessment (TLFB) | Baseline, 1-month follow-up
  Daily cannabis use is assessed using the TLFB method, a validated self-report instrument used to collect retrospective estimates of daily cannabis use.
Change in cannabis withdrawal symptoms, measured by the Cannabis Withdrawal Scale (CWS) | Baseline, 1-month follow-up
  The CWS assesses withdrawal symptoms experienced over the last 24 hours and consists of 19 statements. For each statement, its negative impact on normal daily activities is rated on a likert scale from 0 (not at all) to 10 (extremely). The total score ranges from 0 to 190; higher scores indicate that withdrawal symptoms have a larger negative impact on normal daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and risk of re-identification.